CLINICAL TRIAL: NCT04423484
Title: Therapeutic Recommendations for the Treatment of Children With Nephroblastoma in Africa.
Brief Title: Therapeutic Recommendations for Nephroblastoma
Acronym: GFANEPHRO20
Status: Recruiting | Type: Observational
Sponsor: French Africa Pediatric Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: GFANEPHRO2020
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Nephroblastoma
MeSH Terms: conditions — Wilms Tumor | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with Nephroblastoma: All children coming into the participating units with suspected Nephroblastoma.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Clinical stage, treatment given and observations of toxicity if any, outcome following treatment and follow up.

SUMMARY:
The study is based on results form 2 previous studies carried out by the GFAOP. The aim of this study is to evaluate the capacity of units to follow the recommendations in the protocol.

DETAILED DESCRIPTION:
The study is based on results form 2 previous studies carried out by the GFAOP. This study aims to evaluate the capacity of units to follow the recommendations in the protocol. It will look mainly at treatment compliance and outcome for the children treated. The study will also evaluate the improvement in treatment compliance and reporting. This work will help the group to evaluate future needs in participating units and help us adapt treatment programmes to local conditions.

ELIGIBILITY:
Inclusion Criteria:

Unilateral Nephroblastoma Tumor Not previously treated The general health of the child will permit treatment.

.

Exclusion Criteria:

Bilateral Nephroblastoma tumor Previously treated Disease too advanced Doubt concerning the diagnosis Treatment Refusal

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children with local Nephroblastoma in all participating units
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the number of cases with local disease. | 5 years
  By evaluating the initial clinical reports and later histological reports to confirm the stage and the diagnosis.
Evaluation of the number of cases with stage IV disease. | 5 Years
  By evaluating the initial clinical reports and later histological reports to confirm the stage.
Evaluating the treatment given. | 5 Years
  Comparison of treatment given and recommended treatment.
Evaluating the follow up after treatment. | 5 Years
  How many children alive or dead after treatment

SECONDARY OUTCOMES:
Why has treatment failed | 5 years
  look at precision of reporting by comparing reports (histological and surgical)

CONTACTS AND LOCATIONS:
Overall Officials: Fatou Binetou Ms DIAGNE AKONDE, Dr, Principal Investigator — French Africa Pediatric Oncology Group
Locations (7):
- Centre Hospitalier Universitaire Pédiatrique Charles De Gaulle, Ouagadougou, Burkina Faso
- CHU de Treichville à ABIDJAN, Abidjan, Abidjan Autonomous District, Côte d’Ivoire
- Democratic Republic of the Congo (2):
  - CUK (Cliniques Universitaires de Kinshasa), Kinshasa
  - Cliniques Universitaires de Lubumbashi (CUL), Lubumbashi
- HJRA, Hôpital universitaire Joseph Ravoahangy Andrianavalona, Antananarivo, Madagascar
- CHU Gabriel Touré (HGT), Bamako, Mali
- Hôpital Aristide Le Dantec, Avenue Pasteur, BP 3001, Dakar, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Undecided